CLINICAL TRIAL: NCT01965652
Title: A Randomized Double-blind, Placebo-controlled, Parallel-group, Multicenter, Phase 3 Study to Evaluate the Long-term Safety of Naldemedine for the Treatment of Opioid-induced Constipation in Subjects With Non-malignant Chronic Pain Receiving Opioid Therapy
Brief Title: Long Term Safety of Naldemedine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1326V9235
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Opioid-induced Constipation
Keywords: Opioid Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naldemedine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naldemedine (Experimental): Participants received 0.2 mg naldemedine tablets orally once daily for 52 weeks.
  Interventions: Drug: Naldemedine
- Placebo (Placebo Comparator): Participants received matching placebo tablets orally once daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naldemedine — Naldemedine 0.2 mg tablet taken orally once a day
  Other Names: S-297995; Symproic®
  Arms: Naldemedine
Drug: Placebo — Placebo tablet taken orally once a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the long-term safety of naldemedine for the treatment of constipation due to opioid therapy.

ELIGIBILITY:
Inclusion Criteria

1. Subjects aged 18 to 80 years inclusive at the time of informed consent
2. Subjects must have non-malignant chronic pain treated and must have opioid induced constipation (OIC)
3. Subjects must be treated with a stable opioid regimen at a total daily dose on average of ≥ 30 mg equivalents of oral morphine sulfate
4. Subjects may or may not be on a routine laxative regimen at the time of Screening

Exclusion Criteria

1. Evidence of significant structural abnormalities of the gastrointestinal (GI) tract
2. Evidence of active medical diseases affecting bowel transit
3. History of pelvic disorders that may be a cause of constipation
4. Surgery (except for minor procedures) within 60 days of Screening
5. History of chronic constipation prior to starting analgesic medication or any potential non-opioid cause of bowel dysfunction that may be a major contributor to the constipation (e.g. mechanical GI obstruction)
6. Subjects who have never taken laxatives for the treatment of OIC
7. Current use of any prohibited medication including opioid antagonists, partial or mixed agonists/antagonists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2016-01-12 (Actual); Study Completion 2016-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (186):
- United States (99):
  - Shionogi Research Site, Birmingham, Alabama
  - Shionogi Research Site, Mobile, Alabama
  - Shionogi Research Site, Chandler, Arizona
  - Shionogi Research Site, Glendale, Arizona
  - Shionogi Research Site, Goodyear, Arizona
  - Shionogi Research Site, Mesa, Arizona
  - Shionogi Research Site, Phoenix, Arizona
  - Shionogi Research Site, Tucson, Arizona
  - Shionogi Research Site, Fountain Valley, California
  - Shionogi Research Site, Garden Grove, California
  - Shionogi Research Site, Glendale, California
  - Shionogi Research Site, Long Beach, California
  - Shionogi Research Site, Los Angeles, California
  - Shionogi Research Site, Oceanside, California
  - Shionogi Research Site, Sacramento, California
  - Shionogi Research Site, Santa Ana, California
  - Shionogi Research Site, Upland, California
  - Shionogi Research Site, Colorado Springs, Colorado
  - Shionogi Research Site, Boynton Beach, Florida
  - Shionogi Research Site, Brandon, Florida
  - Shionogi Research Site, Brooksville, Florida
  - Shionogi Research Site, Clearwater, Florida
  - Shionogi Research Site, Fort Myers, Florida
  - Shionogi Research Site, Jacksonville, Florida
  - Shionogi Research Site, Lake City, Florida
  - Shionogi Research Site, Lakeland, Florida
  - Shionogi Research Site, Orlando, Florida
  - Shionogi Research Site, South Miami, Florida
  - Shionogi Research Site, St. Petersburg, Florida
  - Shionogi Research Site, Tampa, Florida
  - Shionogi Research Site, Atlanta, Georgia
  - Shionogi Research Site, Blue Ridge, Georgia
  - Shionogi Research Site, Decatur, Georgia
  - Shionogi Research Site, Savannah, Georgia
  - Shionogi Research Site, Boise, Idaho
  - Shionogi Research Site, Aurora, Illinois
  - Shionogi Research Site, Bloomington, Illinois
  - Shionogi Research Site, Decatur, Illinois
  - Shionogi Research Site, Rockford, Illinois
  - Shionogi Research Site, Schaumburg, Illinois
  - Shionogi Research Site, Evansville, Indiana
  - Shionogi Research Site, Lafayette, Indiana
  - Shionogi Research Site, Valparaiso, Indiana
  - Shionogi Research Site, Augusta, Kansas
  - Shionogi Research Site, Newton, Kansas
  - Shionogi Research Site, Wichita, Kansas
  - Shionogi Research Site, Hartford, Kentucky
  - Shionogi Research Site, Eunice, Louisiana
  - Shionogi Research Site, Lake Charles, Louisiana
  - Shionogi Research Site, Mandeville, Louisiana
  - Shionogi Research Site, Brockton, Massachusetts
  - Shionogi Research Site, Fall River, Massachusetts
  - Shionogi Research Site, New Bedford, Massachusetts
  - Shionogi Research Site, Rochester, Michigan
  - Shionogi Research Site, Saginaw, Michigan
  - Shionogi Research Site, Traverse City, Michigan
  - Shionogi Research Site, Biloxi, Mississippi
  - Shionogi Research Site, Fremont, Nebraska
  - Shionogi Research Site, Omaha, Nebraska
  - Shionogi Research Site, Henderson, Nevada
  - Shionogi Research Site, Las Vegas, Nevada
  - Shionogi Research Site, Trenton, New Jersey
  - Shionogi Research Site, Albuquerque, New Mexico
  - Shionogi Research Site, New York, New York
  - Shionogi Research Site, Greensboro, North Carolina
  - Shionogi Research Site, Wilmington, North Carolina
  - Shionogi Research Site, Winston-Salem, North Carolina
  - Shionogi Research Site, Akron, Ohio
  - Shionogi Research Site, Canton, Ohio
  - Shionogi Research Site, Columbus, Ohio
  - Shionogi Research Site, Groveport, Ohio
  - Shionogi Research Site, Kettering, Ohio
  - Shionogi Research Site, Lebanon, Ohio
  - Shionogi Research Site, Marion, Ohio
  - Shionogi Research Site, Munroe Falls, Ohio
  - Shionogi Research Site, Oklahoma City, Oklahoma
  - Shionogi Research Site, Tulsa, Oklahoma
  - Shionogi Research Site, Portland, Oregon
  - Shionogi Research Site, Huntingdon Valley, Pennsylvania
  - Shionogi Research Site, Jenkintown, Pennsylvania
  - Shionogi Research Site, Lansdale, Pennsylvania
  - Shionogi Research Site, Charleston, South Carolina
  - Shionogi Research Site, Greer, South Carolina
  - Shionogi Research Site, Myrtle Beach, South Carolina
  - Shionogi Research Site, Summerville, South Carolina
  - Shionogi Research Site, Bristol, Tennessee
  - Shionogi Research Site, Milan, Tennessee
  - Shionogi Research Site, Nashville, Tennessee
  - Shionogi Research Site, Austin, Texas
  - Shionogi Research Site, Dallas, Texas
  - Shionogi Research Site, Houston, Texas
  - Shionogi Research Site, Hurst, Texas
  - Shionogi Research Site, Sugar Land, Texas
  - Shionogi Research Site, Bountiful, Utah
  - Shionogi Research Site, Salt Lake City, Utah
  - Shionogi Research Site, South Ogden, Utah
  - Shionogi Research Site, Richmond, Virginia
  - Shionogi Research Site, Bellevue, Washington
  - Shionogi Research Site, Edmonds, Washington
- Australia (9):
  - Shionogi Research Site, Adelaide
  - Shionogi Research Site, Bedford Park
  - Shionogi Research Site, Camperdown
  - Shionogi Research Site, Carina Heights
  - Shionogi Research Site, Caulfield South
  - Shionogi Research Site, Malvern East
  - Shionogi Research Site, Nambour
  - Shionogi Research Site, Sherwood
  - Shionogi Research Site, St Leonards
- Austria (3):
  - Shionogi Research Site, Linz
  - Shionogi Research Site, Vienna
  - Shionogi Research Site, Zams
- Canada (6):
  - Shionogi Research Site, London
  - Shionogi Research Site, Mirabel
  - Shionogi Research Site, Sarnia
  - Shionogi Research Site, Sherbrooke
  - Shionogi Research Site, Toronto
  - Shionogi Research Site, Vancouver
- Czechia (5):
  - Shionogi Research Site, Benešov
  - Shionogi Research Site, Olomouc
  - Shionogi Research Site, Ostrava
  - Shionogi Research Site, Pardubice
  - Shionogi Research Site, Pribram V- Zdabor
- Denmark (3):
  - Shionogi Research Site, Glostrup Municipality
  - Shionogi Research Site, Hellerup
  - Shionogi Research Site, Odense
- Shionogi Research Site, Soulaine Sur Aubance, France
- Germany (11):
  - Shionogi Research Site, Berlin
  - Shionogi Research Site, Dresden
  - Shionogi Research Site, Halle
  - Shionogi Research Site, Hamburg
  - Shionogi Research Site, Hanover
  - Shionogi Research Site, Kassel
  - Shionogi Research Site, Leipzig
  - Shionogi Research Site, Lünen
  - Shionogi Research Site, Mainz
  - Shionogi Research Site, Münster
  - Shionogi Research Site, Stadtroda
- Hungary (5):
  - Shionogi Research Site, Balatonfüred
  - Shionogi Research Site, Budapest
  - Shionogi Research Site, Debrecen
  - Shionogi Research Site, Hatvan
  - Shionogi Research Site, Szikszó
- Israel (4):
  - Shionogi Research Site, Beersheba
  - Shionogi Research Site, Haifa
  - Shionogi Research Site, Tel Aviv
  - Shionogi Research Site, Tel Litwinsky
- Italy (8):
  - Shionogi Research Site, Asti
  - Shionogi Research Site, Catania
  - Shionogi Research Site, Chieti
  - Shionogi Research Site, Florence
  - Shionogi Research Site, Napoli
  - Shionogi Research Site, Rionero in Vulture
  - Shionogi Research Site, Roma
  - Shionogi Research Site, Rome
- Poland (4):
  - Shionogi Research Site, Chorzów
  - Shionogi Research Site, Gdansk
  - Shionogi Research Site, Katowice
  - Shionogi Research Site, Lublin
- South Africa (5):
  - Shionogi Research Site, Alberton
  - Shionogi Research Site, Lyttelton Centurion
  - Shionogi Research Site, Muckleneuk Pretoria
  - Shionogi Research Site, Pretoria West Pretoria
  - Shionogi Research Site, Worcester
- Spain (3):
  - Shionogi Research Site, Barcelona
  - Shionogi Research Site, Girona
  - Shionogi Research Site, Seville
- Sweden (2):
  - Shionogi Research Site, Skene
  - Shionogi Research Site, Stockholm
- United Kingdom (18):
  - Shionogi Research Site, Bath
  - Shionogi Research Site, Belfast
  - Shionogi Research Site, Bexhill on Sea East Sussex
  - Shionogi Research Site, Chesterfield
  - Shionogi Research Site, Chestfield Kent
  - Shionogi Research Site, Daventry Northants
  - Shionogi Research Site, Devon
  - Shionogi Research Site, Epworth Doncaster
  - Shionogi Research Site, Harrogate
  - Shionogi Research Site, Hinckley
  - Shionogi Research Site, Liverpool
  - Shionogi Research Site, Norwich
  - Shionogi Research Site, Oldham
  - Shionogi Research Site, Peterborough
  - Shionogi Research Site, Randalstown, County Antrim
  - Shionogi Research Site, Spiro Close, Pulborough West Sussex
  - Shionogi Research Site, Wellingborough Northamptonshire
  - Shionogi Research Site, York

REFERENCES:
- [Derived] Camilleri M, Hale M, Morlion B, Tack J, Webster L, Wild J. Naldemedine Improves Patient-Reported Outcomes of Opioid-Induced Constipation in Patients with Chronic Non-Cancer Pain in the COMPOSE Phase 3 Studies. J Pain Res. 2021 Jul 16;14:2179-2189. doi: 10.2147/JPR.S282738. eCollection 2021. PMID 34295186
- [Derived] Webster LR, Hale ME, Yamada T, Wild JE. A Renal Impairment Subgroup Analysis of the Safety and Efficacy of Naldemedine for the Treatment of Opioid-Induced Constipation in Patients with Chronic Non-Cancer Pain Receiving Opioid Therapy. J Pain Res. 2020 Mar 24;13:605-612. doi: 10.2147/JPR.S237833. eCollection 2020. PMID 32280263
- [Derived] Wild J, Webster L, Yamada T, Hale M. Safety and Efficacy of Naldemedine for the Treatment of Opioid-Induced Constipation in Patients with Chronic Non-Cancer Pain Receiving Opioid Therapy: A Subgroup Analysis of Patients >/= 65 Years of Age. Drugs Aging. 2020 Apr;37(4):271-279. doi: 10.1007/s40266-020-00753-2. PMID 32086791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 195 clinical sites in North America (Canada and the United States), Europe (Belgium, Denmark, Estonia, France, Germany, Hungary, Poland, Spain, Sweden, and the United Kingdom), and Africa/Asia Pacific (Australia and South Africa)
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive naldemedine or placebo for 52 weeks. Randomization was stratified based on documented opioid use (average total daily dose [TDD] during the 14-consecutive-day qualifying period) as follows:
  * 30 - 100 mg equivalents of oral morphine sulfate.
  * > 100 mg equivalents of oral morphine sulfate.
Groups:
- Placebo: Participants received placebo tablets orally once daily for 52 weeks.
Period: Overall Study
Arm/Group | Naldemedine | Placebo
Started | 623 (Includes two participants who each enrolled at two different sites) | 623 (Includes three participants who each enrolled at two different sites)
Received Treatment | 622 | 623
Completed | 413 | 413
Not Completed | 210 | 210
Not completed — Adverse Event | 40 | 37
Not completed — Withdrawal by Subject | 62 | 69
Not completed — Lost to Follow-up | 53 | 40
Not completed — Protocol Violation | 34 | 38
Not completed — Death | 3 | 4
Not completed — Other - Miscellaneous | 18 | 21
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study drug. Five participants (2 in the naldemedine group and 3 in the placebo group) were excluded due to double enrollment at different sites. One participant in the placebo arm received naldemedine in error and is included in the naldemedine arm for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Naldemedine | Placebo | Total
Number analyzed (Participants) | 621 | 619 | 1240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (11.68) | 52.7 (10.55) | 53.0 (11.13)
Age, Customized [Number; unit: participants]
  < 40 years | 75 | 68 | 143
  ≥ 40 to < 65 years | 445 | 475 | 920
  ≥ 65 years | 101 | 76 | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 383 | 402 | 785
  Male | 238 | 217 | 455
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 42 | 89
  Not Hispanic or Latino | 574 | 577 | 1151
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 7 | 9
  Asian | 5 | 7 | 12
  Black or African American | 120 | 108 | 228
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  White | 492 | 496 | 988
Stratification by Opioid Dose [Number; unit: participants] — Dose of opioid was calculated using maintenance and breakthrough morphine equivalent dose. If any participants were treated with < 30 mg, the participants were counted in the '30-100' group.
  participants
    30-100 mg | 396 | 392 | 788
    > 100 mg | 225 | 227 | 452

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event was defined as any adverse event (AE) that resulted in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life threatening, or require hospitalization were considered an SAE when, based upon appropriate medical judgment, they jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above.
  Adverse drug reactions (ADRs) were defined as adverse events that were considered by the investigator to be definitely, probably, or possibly related to study drug. Serious ADRs were defined as serious AEs considered by the investigator to be definitely, probably, or possibly related to study drug.
Time Frame: From the first dose of study drug up to 14 days after the last dose of study drug (54 weeks).
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 619
participants
  Adverse events | 425 | 446
  Adverse drug reactions | 149 | 121
  AEs leading to discontinuation of study drug | 39 | 36
  Serious adverse events | 60 | 73
  Serious adverse drug reactions | 3 | 6
  SAEs leading to discontinuation of study drug | 7 | 12
  Deaths | 1 | 3

2. Secondary Outcome: Change From Baseline in the Number of Bowel Movements Per Week
Description: Participants monitored their bowel movements and completed a daily bowel habits diary the week prior to study visits (i.e. during Weeks 11, 23, 35, and 51).
Time Frame: Baseline and Weeks 12, 24, 36, and 52
Population: The intent-to-treat population includes all randomized participants. Five participants were excluded due to double enrollment at different sites.
Measure: Least Squares Mean (Standard Error); unit: bowel movements / week
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
bowel movements / week
  Week 12 | 3.70 (0.163) | 2.42 (0.162)
  Week 24 | 3.77 (0.172) | 2.77 (0.172)
  Week 36 | 3.88 (0.180) | 2.88 (0.177)
  Week 52 | 3.92 (0.184) | 2.92 (0.187)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures — The significance level was set at 0.05 (2-sided). The analysis of efficacy endpoints was not adjusted for multiplicity; hence, the p-values are purely nominal. A mixed-effects model repeated measures (MMRM) method was used for the comparisons; The MMRM method included the opioid dose strata as a covariate and treatment group, time, and time-by-treatment group interaction as fixed effects; LS Mean Difference = 1.28, 95% CI 2-sided [0.83 to 1.72], Standard Error of Mean 0.226
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 1.00, 95% CI 2-sided [0.53 to 1.47], Standard Error of Mean 0.240
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 1.01, 95% CI 2-sided [0.52 to 1.50], Standard Error of Mean 0.249
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p = 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 1.00, 95% CI 2-sided [0.49 to 1.51], Standard Error of Mean 0.259

3. Secondary Outcome: Percentage of Participants Meeting Each Criterion of Laxative Use
Description: Participants who were taking stable routine/regular laxatives at Screening were to continue taking the same regimen throughout the study.
  The percentage of participants meeting each of the criteria below are reported:
  1. Participants not on stable laxatives, defined as participants who did not use laxatives from 28 days prior to the Screening Period to the final dose of study drug or who received only rescue laxative. Rescue is defined as any laxative taken for the first time during the Treatment Period.
  1a. Out of participants who were not on stable laxatives, participants who received rescue laxatives.
  2. Participants on stable laxatives, defined as participants who may have had at least one/any stable laxative use reported from 28 days prior to Screening Period to the final dose of study drug.
  2a. Out of participants who were on stable laxatives, participants who received rescue laxatives.
  3. Participants who did not meet criteria 1 or 2.
Time Frame: From 28 days prior to screening until the end of the treatment period (total of 56 weeks)
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
percentage of participants
  1. Participants not on stable laxatives | 30.0 | 29.5
  1a. Who received rescue laxative: number analyzed (Participants) | 186 | 183
  1a. Who received rescue laxative | 7.0 | 13.1
  2. Participants on stable laxatives | 50.2 | 54.0
  2a. Who received rescue laxative: number analyzed (Participants) | 312 | 335
  2a. Who received rescue laxative | 8.0 | 14.0
  3. Other participants | 19.8 | 16.5

4. Secondary Outcome: Change From Baseline in the Overall Score for Patient Assessment of Constipation Symptoms
Description: The Patient Assessment of Constipation Symptom Questionnaire (PAC-SYM) asked participants to rate the severity of 12 constipation symptoms in the last 2 weeks on a scale from 0 (absent) to 4 (very severe). The overall score was calculated as the mean of all 12 items and ranges from 0 (best) to 4 (worst). A negative change from baseline value indicates improvement.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -1.15 (0.036) | -0.81 (0.036)
  Week 12 | -1.11 (0.039) | -0.86 (0.039)
  Week 24 | -1.16 (0.039) | -0.87 (0.039)
  Week 36 | -1.21 (0.040) | -0.85 (0.040)
  Week 52 | -1.22 (0.041) | -0.98 (0.042)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; The mixed-effects model repeated measures (MMRM) method included treatment group, time, and time-by-treatment group interaction as fixed effects; LS Mean Difference = -0.35, 95% CI 2-sided [-0.44 to -0.25], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.25, 95% CI 2-sided [-0.36 to -0.14], Standard Error of Mean 0.055
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.29, 95% CI 2-sided [-0.40 to -0.18], Standard Error of Mean 0.056
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.35, 95% CI 2-sided [-0.47 to -0.24], Standard Error of Mean 0.057
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.24, 95% CI 2-sided [-0.35 to -0.12], Standard Error of Mean 0.059

5. Secondary Outcome: Change From Baseline in the PAC-SYM Abdominal-symptoms Domain Score
Description: The Patient Assessment of Constipation Symptom Questionnaire (PAC-SYM) asked participants to rate the severity of 12 constipation symptoms in the last 2 weeks on a scale from 0 (absent) to 4 (very severe). The abdominal-symptom domain score was calculated as the mean of the following 4 items: abdominal discomfort, abdominal pain, abdominal bloating and stomach cramps.
  A negative change from baseline value indicates improvement in symptoms.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -0.99 (0.038) | -0.79 (0.038)
  Week 12 | -0.93 (0.042) | -0.78 (0.043)
  Week 24 | -0.99 (0.043) | -0.81 (0.043)
  Week 36 | -1.06 (0.043) | -0.78 (0.043)
  Week 52 | -1.07 (0.045) | -0.94 (0.045)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p = 0.0002, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.20, 95% CI 2-sided [-0.31 to -0.10], Standard Error of Mean 0.054
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p = 0.0173, Mixed-effects model repeated meaures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.14, 95% CI 2-sided [-0.26 to -0.03], Standard Error of Mean 0.060
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p = 0.0035, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.18, 95% CI 2-sided [-0.30 to -0.06], Standard Error of Mean 0.061
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.28, 95% CI 2-sided [-0.40 to -0.16], Standard Error of Mean 0.061
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p = 0.0336, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.14, 95% CI 2-sided [-0.26 to -0.01], Standard Error of Mean 0.064

6. Secondary Outcome: Change From Baseline in the PAC-SYM Rectal-symptoms Domain Score
Description: The Patient Assessment of Constipation Symptom Questionnaire (PAC-SYM) asked participants to rate the severity of 12 constipation symptoms in the last 2 weeks on a scale from 0 (absent) to 4 (very severe). The abdominal-symptom domain score was calculated as the mean of the following 3 items: painful bowel movements, rectal burning during or after a bowel movement, and rectal bleeding or tearing during or after a bowel movement. A negative change from baseline value indicates improvement in symptoms.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -1.00 (0.040) | -0.75 (0.040)
  Week 12 | -0.97 (0.044) | -0.81 (0.045)
  Week 24 | -1.02 (0.046) | -0.79 (0.046)
  Week 36 | -1.02 (0.045) | -0.76 (0.045)
  Week 52 | -1.03 (0.046) | -0.87 (0.047)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.25, 95% CI 2-sided [-0.37 to -0.14], Standard Error of Mean 0.057
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p = 0.0114, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.16, 95% CI 2-sided [-0.28 to -0.04], Standard Error of Mean 0.063
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p = 0.0003, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.23, 95% CI 2-sided [-0.36 to -0.11], Standard Error of Mean 0.065
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.25, 95% CI 2-sided [-0.38 to -0.13], Standard Error of Mean 0.064
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p = 0.0119, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.17, 95% CI 2-sided [-0.29 to -0.04], Standard Error of Mean 0.066

7. Secondary Outcome: Change From Baseline in the PAC-SYM Stool-symptoms Domain Score
Description: The Patient Assessment of Constipation Symptom Questionnaire (PAC-SYM) asked participants to rate the severity of 12 constipation symptoms in the last 2 weeks on a scale from 0 (absent) to 4 (very severe). The stool-symptom domain score was calculated as the mean of the following 5 items: incomplete bowel movements, bowel movements that were too hard, bowel movements that were too small, straining or squeezing to try to pass bowel movements, and false-alarm bowel movements.
  A negative change from baseline value indicates improvement in symptoms.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -1.37 (0.045) | -0.86 (0.045)
  Week 12 | -1.34 (0.046) | -0.96 (0.047)
  Week 24 | -1.37 (0.048) | -0.97 (0.048)
  Week 36 | -1.44 (0.050) | -0.96 (0.050)
  Week 52 | -1.45 (0.051) | -1.08 (0.051)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.51, 95% CI 2-sided [-0.64 to -0.39], Standard Error of Mean 0.063
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.38, 95% CI 2-sided [-0.51 to -0.26], Standard Error of Mean 0.066
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.40, 95% CI 2-sided [-0.54 to -0.27], Standard Error of Mean 0.067
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.48, 95% CI 2-sided [-0.62 to -0.34], Standard Error of Mean 0.071
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.37, 95% CI 2-sided [-0.52 to -0.23], Standard Error of Mean 0.072

8. Secondary Outcome: Change From Baseline in the Patient Assessment of Constipation Quality of Life Overall Score
Description: The Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) consists of 28 questions designed to measure the impact constipation has had on participants' daily life during the past 2 weeks.
  Each question was evaluated by the participant on a five-point scale ranging from 0 (not at all or none of the time) to 4 (extremely or all of the time), where higher scores represent poorer quality of life. The overall score was calculated as the mean of all 28 item scores. A negative change from baseline value indicates improvement.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -1.14 (0.033) | -0.75 (0.033)
  Week 12 | -1.19 (0.036) | -0.83 (0.037)
  Week 24 | -1.19 (0.038) | -0.86 (0.038)
  Week 36 | -1.22 (0.039) | -0.82 (0.039)
  Week 52 | -1.24 (0.039) | -0.94 (0.040)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.40, 95% CI 2-sided [-0.49 to -0.30], Standard Error of Mean 0.047
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.36, 95% CI 2-sided [-0.46 to -0.26], Standard Error of Mean 0.051
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.33, 95% CI 2-sided [-0.43 to -0.22], Standard Error of Mean 0.054
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.40, 95% CI 2-sided [-0.50 to -0.29], Standard Error of Mean 0.055
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.31, 95% CI 2-sided [-0.42 to -0.20], Standard Error of Mean 0.056

9. Secondary Outcome: Change From Baseline in the Physical Discomfort Domain of PAC-QOL
Description: The Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) consists of 28 questions designed to measure the impact constipation has had on participants' daily life during the past 2 weeks.
  Each question was evaluated by the participant on a five-point scale ranging from 0 (not at all or none of the time) to 4 (extremely or all of the time), where higher scores represent poorer quality of life. The physical discomfort domain consists of 4 questions related to bloating, feeling heavy, how much of the time participants felt any physical discomfort and how much time they felt the need to open their bowel but were not able to. The physical discomfort score was calculated as the mean of the 4 individual scores. A negative change from baseline value indicates improvement.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -1.33 (0.040) | -0.94 (0.040)
  Week 12 | -1.27 (0.044) | -0.95 (0.045)
  Week 24 | -1.26 (0.046) | -0.98 (0.046)
  Week 36 | -1.28 (0.048) | -0.94 (0.048)
  Week 52 | -1.38 (0.047) | -1.09 (0.047)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.39, 95% CI 2-sided [-0.50 to -0.28], Standard Error of Mean 0.056
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Anaysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.32, 95% CI 2-sided [-0.44 to -0.20], Standard Error of Mean 0.063
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.40 to -0.15], Standard Error of Mean 0.065
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.34, 95% CI 2-sided [-0.48 to -0.21], Standard Error of Mean 0.068
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.28, 95% CI 2-sided [-0.41 to -0.15], Standard Error of Mean 0.067

10. Secondary Outcome: Change From Baseline in the Psychosocial Discomfort Domain of PAC-QOL
Description: The Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) consists of 28 questions designed to measure the impact constipation has had on participants' daily life during the past 2 weeks.
  Each question was evaluated by the participant on a five-point scale ranging from 0 (not at all or none of the time) to 4 (extremely or all of the time), where higher scores represent poorer quality of life. The psychosocial discomfort domain consists of 8 questions related to participants' embarrassment regarding their constipation and effects of constipation on eating habits and appetite.
  The psychosocial discomfort score was calculated as the mean of the 8 individual scores. A negative change from baseline value indicates improvement.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -0.92 (0.036) | -0.69 (0.036)
  Week 12 | -0.96 (0.039) | -0.72 (0.039)
  Week 24 | -0.97 (0.040) | -0.72 (0.040)
  Week 36 | -0.99 (0.042) | -0.68 (0.042)
  Week 52 | -1.00 (0.043) | -0.80 (0.043)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.24, 95% CI 2-sided [-0.34 to -0.14], Standard Error of Mean 0.051
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.24, 95% CI 2-sided [-0.35 to -0.14], Standard Error of Mean 0.055
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.25, 95% CI 2-sided [-0.36 to -0.14], Standard Error of Mean 0.057
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.31, 95% CI 2-sided [-0.43 to -0.19], Standard Error of Mean 0.059
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p = 0.0006, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.21, 95% CI 2-sided [-0.33 to -0.09], Standard Error of Mean 0.061

11. Secondary Outcome: Change From Baseline in the Worries and Concerns Domain of PAC-QOL
Description: The Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) consists of 28 questions designed to measure the impact constipation has had on participants' daily life during the past 2 weeks.
  Each question was evaluated by the participant on a five-point scale ranging from 0 (not at all or none of the time) to 4 (extremely or all of the time), where higher scores represent poorer quality of life. The worries and concerns domain consists of 11 questions related to participants' feelings and concerns about their constipation. The worries and concerns domain score was calculated as the mean of the 11 individual scores. A negative change from baseline value indicates improvement.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -1.14 (0.038) | -0.74 (0.038)
  Week 12 | -1.21 (0.042) | -0.85 (0.042)
  Week 24 | -1.19 (0.043) | -0.87 (0.043)
  Week 36 | -1.23 (0.044) | -0.81 (0.044)
  Week 52 | -1.24 (0.045) | -0.92 (0.045)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.39, 95% CI 2-sided [-0.50 to -0.29], Standard Error of Mean 0.054
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.36, 95% CI 2-sided [-0.48 to -0.24], Standard Error of Mean 0.060
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.33, 95% CI 2-sided [-0.45 to -0.21], Standard Error of Mean 0.061
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.42, 95% CI 2-sided [-0.54 to -0.30], Standard Error of Mean 0.062
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.32, 95% CI 2-sided [-0.44 to -0.19], Standard Error of Mean 0.064

12. Secondary Outcome: Change From Baseline in the Satisfaction Domain of PAC-QOL
Description: The Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) consists of 28 questions designed to measure the impact constipation has had on participants' daily life during the past 2 weeks.
  Each question was evaluated by the participant on a five-point scale ranging from 0 (not at all or none of the time) to 4 (extremely or all of the time), where higher scores represent poorer quality of life. The satisfaction domain consists of 5 questions related to participants' feelings of satisfaction with their bowel function. The satisfaction domain score was calculated as the mean of the 5 individual scores. A negative change from baseline value indicates improvement.
Time Frame: Baseline and Weeks 2, 12, 24, 36, and 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
units on a scale
  Week 2 | -1.37 (0.050) | -0.70 (0.050)
  Week 12 | -1.45 (0.053) | -0.87 (0.053)
  Week 24 | -1.50 (0.054) | -0.99 (0.054)
  Week 36 | -1.53 (0.056) | -1.00 (0.056)
  Week 52 | -1.54 (0.059) | -1.07 (0.059)
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Week 2 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.67, 95% CI 2-sided [-0.81 to -0.53], Standard Error of Mean 0.070
Statistical Analysis 2: Comparison: Naldemedine vs Placebo; Week 12 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.58, 95% CI 2-sided [-0.73 to -0.43], Standard Error of Mean 0.075
Statistical Analysis 3: Comparison: Naldemedine vs Placebo; Week 24 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.51, 95% CI 2-sided [-0.66 to -0.36], Standard Error of Mean 0.077
Statistical Analysis 4: Comparison: Naldemedine vs Placebo; Week 36 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.54, 95% CI 2-sided [-0.69 to -0.38], Standard Error of Mean 0.080
Statistical Analysis 5: Comparison: Naldemedine vs Placebo; Week 52 Analysis; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -0.48, 95% CI 2-sided [-0.64 to -0.32], Standard Error of Mean 0.083

13. Secondary Outcome: Participant Global Satisfaction
Description: Participants were asked to rate their degree of satisfaction of constipation and abdominal symptoms from the start of study drug dosing to Week 52 (or early termination).
  Satisfaction was rated based on the following seven grades:
  * Grade 1 = markedly worsened
  * Grade 2 = moderately worsened
  * Grade 3 = slightly worsened
  * Grade 4 = unchanged
  * Grade 5 = slightly improved
  * Grade 6 = moderately improved
  * Grade 7 = markedly improved
Time Frame: Week 52 or early termination visit
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Naldemedine | Placebo
Number analyzed (Participants) | 621 | 620
percentage of participants
  Markedly worsened | 2.4 | 2.0
  Moderately worsened | 0.6 | 2.8
  Slightly worsened | 1.0 | 2.2
  Unchanged | 14.9 | 33.5
  Slightly improved | 20.1 | 23.0
  Moderately improved | 26.0 | 17.7
  Markedly improved | 35.0 | 18.8
Statistical Analysis 1: Comparison: Naldemedine vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 14 days after the last dose of study drug (54 weeks).
Description: The safety population included all participants who were randomized and received at least 1 dose of study drug and were analyzed by the treatment actually received. Five participants (2 in the naldemedine group and 3 in the placebo group) were excluded due to double enrollment at different sites. One participant in the placebo arm received naldemedine in error and is included in the naldemedine arm for safety analyses.
Arm/Group | Naldemedine | Placebo
Serious Adverse Events (participants affected / at risk) | 60/621 | 73/619
Other Adverse Events (participants affected / at risk) | 225/621 | 179/619
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naldemedine (N=621) | Placebo (N=619)
Appendicitis (Infections and infestations) | 1 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2
Cellulitis Orbital (Infections and infestations) | 0 | 1
Incision Site Infection (Infections and infestations) | 0 | 1
Infected Skin Ulcer (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 1
Localised Infection (Infections and infestations) | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 4
Pneumonia Bacterial (Infections and infestations) | 0 | 1
Post Procedural Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Tooth Abscess (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection Pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Acute Psychosis (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1
Panic Attack (Psychiatric disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 1
Stress (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Cervicobrachial Syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1
Spinal Claudication (Nervous system disorders) | 0 | 1
Toxic Encephalopathy (Nervous system disorders) | 2 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 2 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 2
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 2
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Femoral Artery Occlusion (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Peripheral Vascular Disorder (Vascular disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastric Varices (Gastrointestinal disorders) | 0 | 1
Gastric Volvulus (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder Prolapse (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Sickle Cell Anaemia with Crisis (Congenital, familial and genetic disorders) | 1 | 0
Device Dislocation (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 3
Surgical Failure (General disorders) | 0 | 1
Blood Potassium Increased (Investigations) | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 0 | 1
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naldemedine (N=621) | Placebo (N=619)
Upper Respiratory Tract Infection (Infections and infestations) | 36 | 33
Urinary Tract Infection (Infections and infestations) | 38 | 51
Headache (Nervous system disorders) | 28 | 33
Abdominal Pain (Gastrointestinal disorders) | 50 | 18
Diarrhoea (Gastrointestinal disorders) | 68 | 33
Nausea (Gastrointestinal disorders) | 49 | 35
Vomiting (Gastrointestinal disorders) | 36 | 18
Back Pain (Musculoskeletal and connective tissue disorders) | 34 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.